CLINICAL TRIAL: NCT02886676
Title: Effect of Arthrospira Platensis (Spirulina) as an Adjunct to Scaling and Root Planing on Salivary Antioxidant Levels in Chronic Periodontitis Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tatyasaheb Kore Dental College (Other)
Responsible Party: Principal Investigator, Dr. Pradnya Rajendra Khatavkar, post graduate syudent, Tatyasaheb Kore Dental College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: panu2511
Record Dates: First submitted 2016-08-27; First posted 2016-09-01 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Spirulina capsules and scaling & root planing (Experimental): Patients in test group will be provided with Spirulina capsules 2gm daily, after meals for 1 month
  Interventions: Drug: Spirulina capsules
- Placebo capsules and scaling & root planing (Active Comparator): Patients in test group will be provided with placebo capsules after meals for 1 month
  Interventions: Drug: Spirulina capsules

INTERVENTIONS:
Drug: Spirulina capsules — Spirulina capsules 2gm daily for 1 month

SUMMARY:
Introduction- Oxidative stress plays a causative role in pathogenesis of periodontal disease.

It has been reported that Spirulina platensis or its active ingredient C phycocyanin (CPC) exerts anti-inflammatory, anti-oxidative and inhibitory effects on prostaglandin and leukotriene biosynthesis.

Aim- To evaluate the effect of dietary spirulina as an adjunct to SRP on salivary antioxidants level in CP subjects.

Materials And Methods- The study was a randomized double-blind clinical and biochemical trial in which 70 subjects with CP in the age group of 40-55 years, reporting to Department of Periodontology, TKDC and RC, New Pargaon, were equally and randomly divided into Test Group (TG) and Control Group (CG). TG was given 2 gm Spirulina capsules daily, after meals for 1 month and CG was not given any supplementary diet. SRP was done at baseline in TG and CG. Whole saliva sample was collected. Clinical and biochemical parameters will be recorded at baseline, 1 month & 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with CP (moderate and severe)as per CDC criteria 2007.
2. Patients without any known systemic diseases.

Exclusion Criteria:

1. Patients who have taken anti-inflammatory/antibiotic/antioxidant within 3 months of beginning of study.
2. Subjects who have undergone periodontal treatment within six months of inception of study.
3. Tobacco habits in any form and alcoholics.
4. Pregnant and lactating women.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2015-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Superoxide dismutase (SOD) | 3 month
Malondialdehyde (MDA) | 3 month

SECONDARY OUTCOMES:
plaque index | 3 month
Gingival bleeding index | 3 month
Sulcus bleeding index (SBI) | 3 month
Probing depth (PD) | 3 month
Clinical Attachment Level (CAL) | 3 month